CLINICAL TRIAL: NCT02949973
Title: An Exploratory Study Assessing the Short Term Predictors of Remission of Voclosporin 23.7mg Twice Daily (BID) in Combination With Standard of Care in Patients With Active Lupus Nephritis
Brief Title: Aurinia Early Urinary Protein Reduction Predicts Response
Acronym: AURION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aurinia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUR-VCS-2014-01
Record Dates: First submitted 2016-10-26; First posted 2016-10-31 (Estimated); Results first posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Lupus Nephritis
Keywords: lupus nephritis; calcineurin inhibitors; voclosporin
MeSH Terms: conditions — Lupus Nephritis | interventions — voclosporin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Voclosporin (Experimental): Voclosporin, oral, 23.7 mg twice daily (BID)
  Interventions: Drug: voclosporin

INTERVENTIONS:
Drug: voclosporin
  Other Names: ISA247

SUMMARY:
An exploratory study assessing the ability of biomarkers measured at 8 weeks to predict clinical response over 24 and 48 weeks in subjects taking voclosporin 23.7 mg twice daily (BID) in combination with standard of care in patients with active lupus nephritis

DETAILED DESCRIPTION:
Voclosporin is a novel calcineurin inhibitor (CNI) intended for use in the prevention of organ graft rejection and for the treatment of autoimmune diseases. The aim of the current development program is to investigate whether voclosporin added to the standard of care treatment in active Lupus Nephritis (LN) is able to reduce disease activity, as measured by a reduction in proteinuria. The background therapy will be mycophenolate mofetil (MMF) 2 g daily, initial treatment with IV methylprednisolone followed by a reducing course of oral corticosteroids. Patients with active, flaring LN will be eligible to enter the study. They are required to have a diagnosis of LN according to established diagnostic criteria (American College of Rheumatology) and clinical and biopsy features suggestive of active nephritis. Efficacy will be assessed by the ability of the drug combination to reduce the level of proteinuria while demonstrating an acceptable safety profile.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of systemic lupus erythematosus (SLE) according to the American College of Rheumatology criteria (1997; see Appendix 6).
* Kidney biopsy within 24 months prior to screening with a histologic diagnosis of lupus nephritis International Society of Nephrology/Renal Pathology Society Classes III, IV-S or IV-G, (A) or (A/C); or Class V, alone or in combination with Class III or IV.
* Laboratory evidence of active nephritis at screening, defined as: Class III, IV-S or Class IV-G (proteinuria ≥1000 mg/24 hours when assessed by 24 hour urine collection, defined by a urine protein/creatinine ratio (UPCR) of ≥1.0 mg/mg assessed in a first morning void urine specimen). Class V, alone or in combination with Class III or IV, (proteinuria ≥1,500 mg/24 hours when assessed by 24 hour urine collection, defined by a UPCR of ≥1.5 mg/mg assessed in a first morning void urine specimen).

Key Exclusion Criteria:

* Estimated glomerular filtration rate (eGFR) as calculated by the Chronic Kidney Disease Epidemiology Collaboration equation of ≤45 mL/min/1.73 m2 at screening
* Currently requiring renal dialysis (hemodialysis or peritoneal dialysis) or expected to require dialysis during the study period.
* A previous kidney transplant or planned transplant within study treatment period.
* Malignancy within 5 years of screening, with the exception of basal and squamous cell carcinomas treated by complete excision. Subjects with cervical dysplasia that is cervical intraepithelial neoplasia 1, but have been treated with conization or loop electrosurgical excision procedure, and have had a normal repeat Papanicolaou smear test (PAP) are allowed.
* Lymphoproliferative disease or previous total lymphoid irradiation.
* Severe viral infection (such as Cytomegalovirus (CMV), Hepatitis B virus (HBV), Hepatitis C virus (HCV)) within 3 months of screening; or known human immunodeficiency virus infection.
* Active tuberculosis (TB), or known history of TB/evidence of old TB if not taking prophylaxis with isoniazid.
* Other known clinically significant active medical conditions, such as:
* Severe cardiovascular disease including congestive heart failure, history of cardiac dysrhythmia or congenital long QT syndrome. QT interval duration corrected for heart rate using method of Fridericia (QTcF) exceeding 480 msec in the presence of a normal QRS interval (<110 msec) at time of screening will result in exclusion.
* Liver dysfunction (aspartate aminotransferase, alanine aminotransferase, or bilirubin greater than 2.5 times the upper limit of normal) at screening and confirmed before enrollment.
* Chronic obstructive pulmonary disease or asthma requiring oral steroids.
* Bone marrow insufficiency unrelated to active systemic lupus erythematosus (SLE) (according to Investigator judgment) with white blood cell count <2,500/mm3; absolute neutrophil count <1.3 × 103/μL; thrombocytopenia (platelet count <50,000/mm3).
* Active bleeding disorders.
* Current infection requiring IV antibiotics.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2017-02-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- AURION Site, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Voclosporin 23.7 mg Twice Daily (BID) in Combination With Standard of Care: Voclosporin 23.7 mg twice daily (BID)
Period: Overall Study
Arm/Group | Voclosporin 23.7 mg Twice Daily (BID) in Combination With Standard of Care
Started | 10
Completed | 9
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Voclosporin 23.7 mg Twice Daily (BID) in Combination With Standard of Care
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] — Safety Population
  years | 28.7 (5.14)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety Population
  Participants
    Female | 10
    Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Safety Population
  Participants
    American Indian or Alaska Native | 0
    Asian | 10
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Malaysia | 10
Duration of systemic lupus erythematosus, proteinuria and lupus nephritis [Mean (Standard Deviation); unit: years]
  Duration of systemic lupus erythematosus (SLE) | 7.3 (3.23)
  Duration of proteinuria | 5.9 (3.38)
  Duration of Lupus Nephritis (LN) | 5.8 (3.49)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reduction or Normalization of Urine Protein/Creatinine Ratio (UPCR)
Time Frame: 24 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin 23.7 mg Twice Daily (BID) in Combination With Standard of Care
Number analyzed (Participants) | 10
Participants | 7
Statistical Analysis 1: Comparison: Voclosporin 23.7 mg Twice Daily (BID) in Combination With Standard of Care; Test type: Other; Percentage = 70

2. Primary Outcome: Number of Participants With Reduction or Normalization of Anti ds DNA
Time Frame: 24 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin 23.7 mg Twice Daily (BID) in Combination With Standard of Care
Number analyzed (Participants) | 10
Participants | 4
Statistical Analysis 1: Comparison: Voclosporin 23.7 mg Twice Daily (BID) in Combination With Standard of Care; Test type: Other; Percentage = 40

3. Primary Outcome: Number of Participants With Reduction or Normalization of C3
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin 23.7 mg Twice Daily (BID) in Combination With Standard of Care
Number analyzed (Participants) | 10
Participants | 2
Statistical Analysis 1: Comparison: Voclosporin 23.7 mg Twice Daily (BID) in Combination With Standard of Care; Test type: Other; Percentage = 20

4. Primary Outcome: Number of Participants With Reduction or Normalization of C4
Time Frame: 24 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin 23.7 mg Twice Daily (BID) in Combination With Standard of Care
Number analyzed (Participants) | 10
Participants | 2
Statistical Analysis 1: Comparison: Voclosporin 23.7 mg Twice Daily (BID) in Combination With Standard of Care; Test type: Other; Percentage = 20

5. Secondary Outcome: Number of Participants With Complete Remission at Week 24
Description: * Confirmed Protein/creatinine ratio of ≤0.5 mg/mg and
  * eGFR ≥ 60 mL/min/1.73 m2 or no confirmed decrease from baseline in eGFR of ≥20%
Time Frame: week 24
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin 23.7 mg Twice Daily (BID) in Combination With Standard of Care
Number analyzed (Participants) | 10
Participants | 7
Statistical Analysis 1: Comparison: Voclosporin 23.7 mg Twice Daily (BID) in Combination With Standard of Care; Test type: Other; Percentage = 70, 95% CI 2-sided [34.8 to 93.3]

6. Secondary Outcome: Number of Participants With Complete Remission at Week 48
Description: * Confirmed Protein/creatinine ratio of ≤0.5 mg/mg and
  * eGFR ≥ 60 mL/min/1.73 m2 or no confirmed decrease from baseline in eGFR of ≥20%
  Safety Population - 2 subjects failed to provide sufficient data to ascertain week 48 response
Time Frame: week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin 23.7 mg Twice Daily (BID) in Combination With Standard of Care
Number analyzed (Participants) | 8
Participants | 4
Statistical Analysis 1: Comparison: Voclosporin 23.7 mg Twice Daily (BID) in Combination With Standard of Care; Test type: Other; Percentage = 50, 95% CI 2-sided [15.7 to 84.3]

ADVERSE EVENTS:
Arm/Group | Voclosporin 23.7 mg Twice Daily (BID) in Combination With Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Voclosporin 23.7 mg Twice Daily (BID) in Combination With Standard of Care (N=10)
Acute Tonsilitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Voclosporin 23.7 mg Twice Daily (BID) in Combination With Standard of Care (N=10)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Otorrhoea (Ear and labyrinth disorders) | 1 (2)
Cushingoid (Endocrine disorders) | 1 (1)
Chalazion (Eye disorders) | 1 (1)
Conjunctival Haemorrhage (Eye disorders) | 1 (1)
Eyelid Oedema (Eye disorders) | 1 (1)
Vision Blurred (Eye disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (6)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Gingival Bleeding (Gastrointestinal disorders) | 1 (1)
Gingival Pain (Gastrointestinal disorders) | 1 (1)
Gingival Swelling (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Tongue Ulceration (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Chest Pain (General disorders) | 2 (2)
Local Swelling (General disorders) | 2 (2)
Oedema (General disorders) | 2 (2)
Oedema Peripheral (General disorders) | 1 (2)
Pyrexia (General disorders) | 5 (10)
Herpes Zoster (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2)
Tonsillitis (Infections and infestations) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (7)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Viral Pharyngitis (Infections and infestations) | 1 (1)
Breath Sounds Abnormal (Investigations) | 1 (1)
Glomerular Filtration Rate Decreased (Investigations) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Burning Sensation (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3)
Headache (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1)
Menstruation Irregular (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Hirsutism (Skin and subcutaneous tissue disorders) | 1 (1)
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Rash Macular (Skin and subcutaneous tissue disorders) | 1 (1)
Rash Papular (Skin and subcutaneous tissue disorders) | 1 (1)
Swelling Face (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No